CLINICAL TRIAL: NCT05744427
Title: Phase I/II Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of JSKN003 in Chinese Subjects With Advanced Solid Tumors
Brief Title: Safety and Tolerability of JSKN003 in Chinese Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JSKN003-102
Record Dates: First submitted 2023-01-10; First posted 2023-02-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Dose escalation and expansion period (Experimental): in dose escalation and expansion period，total 8 dose groups were designed. Subjects will be give dose 1.0, 2.1, 4.2, 5.2, 6.3, 7.3, 8.4 and 10.5 mg/kg Q3W based on DLT results.
  Interventions: Drug: JSKN003
- cohort 1 in phase II (Experimental)
  Interventions: Drug: JSKN003
- cohort 2 in phase II (Experimental)
  Interventions: Drug: JSKN003
- cohort 3 in phase II (Experimental)
  Interventions: Drug: JSKN003
- cohort 4 in phase II (Experimental)
  Interventions: Drug: JSKN003
- cohort 5 in phase II (Experimental)
  Interventions: Drug: JSKN003
- cohort 6 in phase II (Experimental)
  Interventions: Drug: JSKN003
- cohort 7 in phase II (Experimental)
  Interventions: Drug: JSKN003

INTERVENTIONS:
Drug: JSKN003 — JSKN003 should be administered intravenously on the first day of each 3-week cycle.

SUMMARY:
This is an open, multicenter study of phase I/II in Chinese subjects with unresectable locally advanced/metastatic solid tumors. It is divided into the dose escalation period and the cohort expansion period. A total of 8 dose groups (Q3W on the first day of intravenous administration) were designed in the dose escalation period. The initial dose was 1.0mg/kg administered Q3W, with a DLT observation period of 21 days. In the dose expansion phase, 7 cohorts were established.

DETAILED DESCRIPTION:
A total of eight dose groups (Q3W, intravenous administration on the first day of each cycle) were designed in the dose escalation period. The dose groups were 1.0, 2.1, 4.2, 5.2, 6.3, 7.3, 8.4 and 10.5 mg/kg. The BOIN design, incorporating accelerated titration, was used, and the DLT observation period was set at 21 days.

The specific steps for implementing the BOIN design in the clinical trial are as follows:

1. Perform the accelerated titration as follows: Assign the first patient to dose level 1. If this patient does not develop dose-limiting toxicity (DLT), the second patient will be treated at the next higher dose level. Treat one patient at a time and continue the dose-escalation process until the first DLT is observed, or a second grade 2 toxicity occurs, or the highest dose is reached. Two more patients were then treated on the current dose. After that, follow steps 2 and 3 and take the number of cases in each group as 3 to treat the follow-up patients.
2. Assign the dose to the next group of subjects according to the dose rise and fall rule shown in the Bayesian Optimal interval (BOIN) decision table.
3. Repeat Step 2 until the set maximum sample size of 45 or the number of evaluable subjects treated at the current dose reaches 12 and the current decision is to maintain the current dose according to the rise and fall rule of the dose rise and fall decision table.

After the dose escalation period was completed, order preserving regression was used to determine MTD. This calculation can be achieved by "Select MTD" in BOIN online software (Zhou et al., 2020). Specifically, the dose whose toxicity rate is closest to the target toxicity rate estimated by isotropic regression is identified as the MTD. During the dose escalation period, the sponsor may, with the approval of the SMC, expand in the appropriate dose group based on the safety, efficacy and external data obtained during the dose escalation period, as long as the number of patients in the extended dose group is consistent with the total sample size during the dose expansion period. Safety monitoring can still be conducted based on the exclusion boundary in the decision table during dose expansion. The patient data of the extended dose group were not involved in the up-down dose decision and the isotonic regression calculation during the dose escalation period.

The Safety Monitoring Committee (SMC) will perform ongoing safety assessment during the dose escalation period. The safety data of each dose group should be reviewed and approved by the SMC before initiating the administration of the next dose group. If additional safety, efficacy, and PK data are required for a dose group by SMC resolution, subjects may continue enrollment in this dose group after completing the BOIN dose eescalation; If the SMC has decided that a dose group can proceed to the cohort extension phase, it is permitted to proceed directly to the cohort extension phase in that dose group. The composition and responsibilities of the SMC will be further detailed in the SMC Constitution.

The recommended dose for cohort expansion (RDE) will be determined by the SMC based on safety/tolerability, PK data, and preliminary antitumor activity, as well as other available data. RDE can be at or below the MTD; RDE may also vary for different indications.

The SMC and sponsor will evaluate the validity of the maximum tolerated dose (MTD) determined by the BOIN design based on data from clinical studies of dose escalation and dose extension, and determine whether it is necessary to explore the higher dose group of 12.6 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old, male or female, and willing to follow the study procedure on the date of signing the informed consent;
2. ECOG score 0 or 1, expected survival ≥12 weeks;
3. Unresectable locally advanced or metastatic solid tumors with pathologic documented confirmation.
4. Measurable lesions at baseline according to RECIST 1.1 criteria; If the subject has only one measurable lesion at baseline, the lesion area must not have received prior radiotherapy or there is evidence of significant progression after the end of radiotherapy.
5. Agrees to provide adequate paraffin sections or fresh tissue specimens of the tumor for testing;
6. Laboratory tests within 7 days or cardiac ultrasound within 28 days prior to the first dose meet the protocol criteria.
7. Adequate washout from prior therapy prior to the first dose.
8. A fertile female subject or a fertile male subject with fertile partner agrees to use highly effective contraception (annual failure rate less than 1%) from the time of initial dosing to 180 days after the end of dosing. Pregnancy test results must be negative for fertile female subjects within 7 days prior to initial administration (fertile women are defined as premenopausal women with no recorded tubal ligation or hysterectomy, or women who have been menopausal for less than 1 year);

Exclusion Criteria:

1. Subjects with untreated active brain metastases or meningeal metastases;
2. History of other primary malignant tumors;
3. Previously received topoisomerase I inhibitor antibody conjugate drug;
4. Has uncontrolled comorbidities as specified by the protocol；
5. Past or current history of interstitial pneumonia/lung disease requiring systemic hormonal therapy, or suspected interstitial pneumonia/lung disease that cannot be ruled out by imaging during screening;
6. Subjects with uncontrolled large serous cavity effusion or moderate to large serous cavity effusion requiring repeated drainage (recurrent within 2 weeks after intervention) such as pleural effusion, pericardial effusion, ascites, etc.;
7. Toxicity from previous antitumor therapy has not resolved to Grade 1 or lower as defined by NCI-CTCAE v5.0.
8. Systemic corticosteroids (≥10 mg/ day of prednisone, or equivalent of other corticosteroids) or immunosuppressant therapy were required within 14 days prior to initial administration in this study;
9. Has a history of life-threatening anaphylaxis or known hypersensitivity to any component or excipient in the JSKN003 drug formulation.
10. History of trastuzumab-induced anaphylaxis (Grade ≥3), angioedema, or severe hypotension.
11. Subjects with gastrointestinal tumors who are known to have lost 10% or more of their body weight within three months prior to signing the informed consent form.
12. Other conditions that the investigator considers unsuitable to participate in this clinical trial, including but not limited to psychiatric disorders, alcoholism or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT (dose escalation period) in phase 1. | Up to 12 months
  Incidence of dose-limiting toxicity (DLT) in the dose escalation period
Maximum Tolerated Dose (MTD) or RP2D in phase 1。 | Up to 12 months
  MTD (Maximum tolerated Dose) is the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate based on the BOIN Design
Percentage of Participants Experiencing Any Treatment Emergent Adverse Events and Serious Treatment Emergent Adverse Events in phase 1. | Throughout the duration of the study, approximately 2 years
  TEAE and SAE were graded according to CTCAE 5.0
Objective Response Rate (ORR) in phase 2 | Throughout the duration of the study, approximately 2 years
  Objective response rate (ORR) was defined as the proportion of participants who achieve either complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST v1.1）

SECONDARY OUTCOMES:
Clinical benefit rates (CBR) | Throughout the duration of the study, approximately 2 years
  Clinical benefit rate (CR+PR+[stable disease (SD) ≥ 6 months]) is defined as those participants with best response as CR or PR or else SD with a duration of at least 6 months. SD for 6 months duration was defined as the time from the first dose to the first documentation of PD or to the last adequate response assessment prior to data cut-off date, whichever is earlier.
Progression Free Survival (PFS) | Throughout the duration of the study, approximately 2 years
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death from any cause
Cmax of JSKN003 | Throughout the duration of the study, approximately 2 years
  Maximum (Peak) observed blood concentration (Cmax) of JSKN003 Following First Dose
Tmax of JSKN003 | Throughout the duration of the study, approximately 2 years
  Time of maximum blood concentration (Tmax) of JSKN003 Following First Dose
AUC of JSKN003 | Throughout the duration of the study, approximately 2 years
  The blood PK parameters of JSKN003 and its analytes for area under the concentration-versus-time curve from time 0 to the last quantifiable concentration as calculated by the linear-up log-down trapezoidal method (AUClast) and AUC from time 0 to infinity (AUCinf) elimination rate constant associated with the terminal phase were estimated using standard non-compartmental methods.
Terminal Elimination Half-life (t1/2) | Throughout the duration of the study, approximately 2 years
  The blood PK parameters of Terminal elimination half-life for JSKN003
Anti-JSKN003 antibody | Throughout the duration of the study, approximately 2 years
  Status (positive or negative) and serum titers of anti-JSKN003 antibody
Duration Of Response (DOR) | Throughout the duration of the study, approximately 2 years
  Defined as the time from the first evaluation of objective response to the first evaluation of PD or death from any cause prior to PD

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, Principal Investigator — Fudan University; Jian Zhang, Principal Investigator — Fudan University
Locations (34):
- China (34):
  - Beijing Cancer Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Sun Yat-sen University Cancer Prevention Center, Guangzhou
  - Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Affiliated Cancer Hospital of Harbin Medical University, Ha’erbin
  - Anhui Provincal Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Linyi City Cancer Hospital, Linyi
  - Linyi City People's Hospital, Linyi
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Gulou Hospital Affiliated to Nanjing University School of Medicine, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Provincial People's Hospital, Nanjing
  - The First Affiliated Hospital of Nanjing Medical University/Jiangsu Provincial People's Hospital, Nanjing
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning
  - Nantong Cancer Hospital, Nantong
  - Affiliated Hospital of Qingdao University, Qingdao
  - Affiliated Cancer Hospital of Fudan University, Shanghai
  - Changhai Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai East Hospital, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Xuzhou Central Hospital, Xuzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou